CLINICAL TRIAL: NCT03439735
Title: Prospective Evaluation of Determinants of Resistance to Endocrine Therapy and a Cyclin-dependent Kinases 4 and 6 (CDK4/6) Inhibitor in Hormone Receptor (HR) Positive Metastatic Breast Cancer (MBC)
Brief Title: Determinants of Resistance to Endocrine Therapy and a Cyclin-dependent Kinases 4 and 6 (CDK4/6) Inhibitor for HR+ MBC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Safeway Foundation (Unknown); Biovica International AB (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J17118; IRB00143030 (Other: JHM-IRB)
Record Dates: First submitted 2017-12-08; First posted 2018-02-20 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic Breast Cancer; Aromatase Inhibitors; Palbociclib; Hormone Receptor Positive Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A: Participants with untreated metastatic disease receiving ET and a CDK 4/6 (Experimental): Participants will undergo blood collection (intervention) at time of initiating treatment with endocrine therapy and palbociclib, at 4 weeks after initiating this treatment, and every 3-4 months while on treatment. If a participant progresses on this treatment, they will have a blood collection at that time.
  Interventions: Drug: Endocrine Therapy and a CDK 4/6 inhibitor
- Cohort B: Participants initiating a CDK 4/6 i after progression on ET. (Experimental): Participants will undergo blood collection (intervention) at time of initiating treatment with endocrine therapy and palbociclib, at 4 weeks after initiating this treatment, and every 3-4 months while on treatment. If a participant progresses on this treatment, they will have a blood collection at that time.
  Interventions: Drug: Endocrine Therapy and a CDK 4/6 inhibitor

INTERVENTIONS:
Drug: Endocrine Therapy and a CDK 4/6 inhibitor — Participants with untreated metastatic disease receiving ET and a CDK 4/6 i as first line therapy.
  Other Names: ET and CDK4/6i
Drug: Endocrine Therapy and a CDK 4/6 inhibitor — Participants initiating a CDK 4/6 i after progression on ET.
  Other Names: ET and CDK4/6i

SUMMARY:
The goal of this research study is to determine if the investigators can predict which participants will respond to endocrine therapy and a cyclin-dependent kinases 4 and 6 (CDK4/6) inhibitor for metastatic breast cancer and which participants will not. Investigators will use information from the tumor tissue and serial blood samples. Investigators hope that a deeper understanding of which participants will respond to this combination and how resistance emerges will allow the investigators to better tailor therapies for metastatic breast cancer.

Subjects will have archived tissue or new biopsy collected at study enrollment. This tissue will undergo special molecular testing. Subjects will also have blood collected at study enrollment and periodically thereafter. This blood will also undergo special molecular testing. Information from this testing will not be available to subjects or their treating physicians as the investigators do not know how this information should impact treatment.

The investigators will collect information about which treatment the subjects receive and how their cancer responds.

Any man or woman being seen at Johns Hopkins for treatment of newly diagnosed estrogen receptor positive (ER+) and/or progesterone receptor positive (PR+) metastatic breast cancer may be eligible.

DETAILED DESCRIPTION:
Resistance to endocrine therapy (ET) invariably develops in patients with estrogen and/or progesterone receptor (ER/ PR) positive metastatic breast cancer (MBC). Data regarding primary resistance and patterns of emergence of acquired resistance in patients treated with endocrine therapy (ET) and cyclin dependent kinase 4 and 6 (CDK4/6) inhibitors are limited. Understanding these mechanisms could result in improved selection of treatment options and provide new targets for therapy development. In this study, we aim to identify and characterize determinants of intrinsic and acquired resistance to endocrine therapy in patients with hormone receptor (HR) positive, human epidermal growth factor receptor 2 (HER2) negative MBC treated with the combination of endocrine therapy (aromatase inhibitor or fulvestrant) and a CDK4/6 inhibitor.

Investigators will determine the prevalence of genomic alterations at baseline in the primary tumor, metastatic tissue and plasma tumor DNA (ptDNA), including in the gene encoding estrogen receptor- alpha (ESR1). The mutational tumor burden in the primary tumor, metastatic tumor and blood will be assessed. Blood samples will be collected at several time points, allowing the detection of changes in molecular markers over time. We will further characterize tissue markers associated with progression and duration of response by evaluating these markers in available tissue obtained at progression. Investigators goal is to evaluate the prevalence and role of known alterations determining endocrine resistance in patients with metastatic disease, as knowledge regarding this population remains limited.The investigators also hope to unveil novel markers of endocrine resistance.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Metastatic (stage IV) breast cancer or locally advanced breast cancer
* Estrogen Receptor (ER) and/or Progesterone Receptor (PR) positive, HER2- negative
* Treatment naïve in metastatic or locally advanced setting and planning to undergo treatment with endocrine therapy (ET) and palbociclib OR receiving first-line ET and palbociclib for metastatic or locally advanced disease.
* Premenopausal women and men must be treated with concurrent luteinizing hormone-releasing hormone (LHRH) agonist as would be standard-of-care.
* Evaluable or measurable disease.
* Tissue from a metastatic site must be available within past 6 months prior to therapy initiation.
* Ability to give voluntary informed consent

Exclusion Criteria:

* Any pregnant or nursing woman
* No history of another primary malignancy within past 5 years. Patients with prior history of in situ cancer or basal or localized squamous cell skin cancer are eligible.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Genetic Mutation | 2 years
  The number of participants who have an ESR1 mutation prior to receiving endocrine therapy and palbociclib.

SECONDARY OUTCOMES:
Genetic Mutation | 4 years
  The amount of time from receiving palbociclib and endocrine therapy to the first detectable ESR1 mutation
Genetic Mutation | 3 years
  Percentage of participants with an ESR1 mutation at the time of progression for those who received treatment with endocrine therapy and palbociclib.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Tao, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No